CLINICAL TRIAL: NCT02403778
Title: Ipilimumab and All-Trans Retinoic Acid Combination Treatment of Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-0948.cc
Record Dates: First submitted 2015-02-23; First posted 2015-03-31 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Melanoma
Keywords: Melanoma; Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Tretinoin; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ipilimumab (Active Comparator): Arm A (No VESANOIDTherapy) will receive the standard of care treatment with ipilimumab only, receiving the standard 4 doses of either 3 or 10 mg/kg ipilimumab every 3 weeks.
  Interventions: Drug: Ipilimumab
- VESANOID (Experimental): Arm B (VESANOID Therapy) will receive the standard 4 doses of either 3 or 10 mg/kg ipilimumab every three weeks plus the supplemental treatment of 150 mg/m2 of VESANOID orally for 3 days surrounding each dose of ipilimumab (day -1, day 0, day +1) for a total of 12 days of VESANOID treatment.
  Interventions: Drug: VESANOID; Drug: Ipilimumab

INTERVENTIONS:
Drug: VESANOID — All-trans retinoic acid (ATRA) is a vitamin A derivative that binds the retinoic acid receptor on MDSCs and differentiates immature monocytes into more mature dendritic cells (12). VESANOID is a standard treatment for patients with acute promyelocytic leukemia (APL).
  Other Names: ATRA; Tretinoin
  Arms: VESANOID
Drug: Ipilimumab — Ipilimumab is current standard of care treatment for melanoma.
  Other Names: IPI

SUMMARY:
The purpose of this study is to assess the safety and efficacy of combined treatment with Ipilimumab and all-trans retinoic acid (ATRA) in melanoma patients.

DETAILED DESCRIPTION:
The successful treatment of melanoma with immune checkpoint inhibitors, such as anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) and Programmed cell death protein 1 (PD-1) antibodies, has altered our thinking and approach to immunotherapy for solid tumors. Despite these advances, only a portion of patients experience a durable response suggesting that there is room for improvement via enhanced immunomodulatory approaches. Anti-CTLA-4 (Ipilimumab) significantly improves overall survival and achieves long-lasting complete responses in some melanoma patients, the number of patients that achieve durable clinical benefit is limited and could be improved by a combined immunomodulatory approach. The objectives of this study are to assess the safety and efficacy of combined treatment with Ipilimumab and all-trans retinoic acid (ATRA) in melanoma patients. We hypothesize that combined treatment with Ipilimumab and ATRA will improve patient responses, increase tumor antigen-specific T cell responses, and decrease immunosuppressive myeloid-derived suppressor cells (MDSCs) in melanoma patients compared to patients treated with Ipilimumab alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 year.
* Patients diagnosed with advanced melanoma.
* Patients that are considered candidates for ipilimumab therapy.
* Patients able to understand and willing to sign a written informed consent documents.
* Patients willing to have regular blood draws, one before treatment and four during or after treatment.

Exclusion Criteria:

* Patients under the age of 18.
* Patients with Stage I or II, melanoma who are not candidates for Ipilimumab.
* Patients that have received systemic treatments within four weeks prior to the beginning of treatment.
* Women that are pregnant or nursing.
* Patients taking immunosuppressive medications.
* Patients with active autoimmune disease.
* Patients with known sensitivity to retinoic acid derivatives.
* Patients with aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin > 2.5 × ULN.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin McCarter, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tobin RP, Jordan KR, Robinson WA, Davis D, Borges VF, Gonzalez R, Lewis KD, McCarter MD. Targeting myeloid-derived suppressor cells using all-trans retinoic acid in melanoma patients treated with Ipilimumab. Int Immunopharmacol. 2018 Oct;63:282-291. doi: 10.1016/j.intimp.2018.08.007. Epub 2018 Aug 16. PMID 30121453

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ipilimumab | VESANOID
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab | VESANOID | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 54.8 [48.2 to 60.1] | 50.4 [33.8 to 66.6] | 52.1 [33.8 to 66.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Safety and tolerability of ipilimumab and VESANOID combination therapy in advanced melanoma patients will be established using the Bayesian approach.
Time Frame: Up to 2 years from the time of study enrollment for each patient.
Measure: Number; unit: Number of events in treatment group
Arm/Group | Ipilimumab | VESANOID
Number analyzed (Participants) | 6 | 4
Number of events in treatment group | 51 | 45

2. Primary Outcome: MDSC Frequency
Description: The frequency of circulating MDSCs will be measured by flow cytometry and calculated as a percentage of the total myeloid cell population. This outcome will be measured at the final study blood draw between 84 and 130 days following the first treatment.
Time Frame: 84 and 130 days following the first treatment
Measure: Mean (Standard Error); unit: % MDSCs of Myeloid Cells
Arm/Group | Ipilimumab | VESANOID
Number analyzed (Participants) | 6 | 4
% MDSCs of Myeloid Cells | 34.35 (6.24) | 7.29 (2.49)

3. Primary Outcome: MDSC Suppressive Function
Description: MDSC suppressive function in peripheral blood will be measured through the activation and proliferation of T cells in the presence of isolated MDSCs. Functional assays will be performed to assess the ability of isolated MDSCs to suppress T-cell responses.
Time Frame: 4 weeks prior to start, Midway thru and at least 30 days post final infusion
Measure: Mean (Standard Deviation); unit: Percentage of Proliferating T Cells
Arm/Group | Ipilimumab | VESANOID
Number analyzed (Participants) | 6 | 4
Percentage of Proliferating T Cells | NA (NA) — Assay not indicative of function no T cell proliferation in controls. | NA (NA) — Assay not indicative of function no T cell proliferation in controls.

4. Secondary Outcome: Changes in the Frequency of Tumor-specific T Cell Responses
Description: Changes in the frequency of tumor-specific T cell responses attributable to the addition of VESANOID to standard ipilimumab therapy will be determined by the frequency of Interferons (IFN)-gamma producing cells after stimulation with melanoma antigens.
Time Frame: 4 weeks prior to start, Midway thru and at least 30 days post final infusion
Measure: Mean (Standard Deviation); unit: Percentage of Activated CD8+ T cells
Arm/Group | Ipilimumab | VESANOID
Number analyzed (Participants) | 6 | 4
Percentage of Activated CD8+ T cells | 6.0975 (4.144) | 14.2833 (7.2221)

5. Secondary Outcome: Unresectable Stage III and STAGE IV
Description: Subjects will be followed for evidence of disease progression.
Time Frame: Up to 2 years from the time of study enrollment for each patient.
Measure: Median (Full Range); unit: Days
Arm/Group | Ipilimumab | VESANOID
Number analyzed (Participants) | 6 | 4
Days | 776 [258 to 912] | 662 [566 to 758]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for up to 2 years from the time of study enrollment for each patient.
Arm/Group | Ipilimumab | VESANOID
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab (N=6) | VESANOID (N=4)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Pseudotumor Cerebri (Nervous system disorders) | 0 (0) | 1 (1)
Colitis or Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Autoimmune Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Elevated ALT (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=6) | VESANOID (N=4)
Colitis (Gastrointestinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 4
Fever (Immune system disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 4
Abdominal Pain (General disorders) | 2 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1
Arthralgias (Immune system disorders) | 0 | 1
Back Pain (General disorders) | 1 | 0
Blurred Vision (Eye disorders) | 0 | 1
Body Aches (increasing) (General disorders) | 0 | 1
Decreased Appetite (General disorders) | 2 | 0
Dry Mouth (General disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 1
Elevated ALT (Hepatobiliary disorders) | 2 | 0
Elevated AST (Hepatobiliary disorders) | 2 | 0
Elevated LFT (Hepatobiliary disorders) | 2 | 1
Erythematous Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Eye Crossing (Eye disorders) | 0 | 1
Facial Flushing (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 2
Malaise (increasing) (General disorders) | 0 | 1
Generalized Flushing (General disorders) | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 1
Itching Eyes (Eye disorders) | 0 | 1
Itching Mouth (General disorders) | 0 | 1
Muscle Ache (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (General disorders) | 0 | 1
Nausea (General disorders) | 4 | 1
Photophobia (Eye disorders) | 0 | 2
Pruritic Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Redness of the Eyes (Eye disorders) | 0 | 1
Skin Color Change (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Peeling (Skin and subcutaneous tissue disorders) | 0 | 1
Uveitis/Iritis (Eye disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02403778/Prot_SAP_000.pdf